CLINICAL TRIAL: NCT01313845
Title: Randomized Double-blind Placebo-controlled Trial of Intravenous Amantadine on Gait Freezing in Patients With Parkinson's Disease
Brief Title: Effect of Intravenous Amantadine on Gait Freezing in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jee-Young Lee (Other)
Collaborators: Seoul National University Boramae Hospital (Other); Samsung Medical Center (Other); Seoul National University Bundang Hospital (Other); Hanyang University (Other)
Responsible Party: Sponsor-Investigator, Jee-Young Lee, assistant professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB11F001
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Amantadine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- amantadine (Active Comparator): administration of intravenous amantadine sulfate 200mg/500ml/bottle 1 bottle infusion over 3 hours, twice a day for consecutive 5 days
  Interventions: Drug: amantadine sulfate
- placebo (Placebo Comparator): administration of 0.9% sodium chloride 500ml/bottle 1 bottle infusion over 3 hours twice a day for consecutive 5 days
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: amantadine sulfate — infusion of amantadine sulfate 100mg/500ml/bottle over 3 hours twice a day
  Other Names: PK-merz
  Arms: amantadine
Drug: 0.9% sodium chloride — infusion of normal saline 500ml/bottle over 3 hours twice a day
  Other Names: normal saline
  Arms: placebo

SUMMARY:
A double-blinded randomized placebo-controlled trial of intravenous amantadine on gait freezing refractory to oral anti-parkinsonian medications in patients with Parkinson's disease.

* administration of IV amantadine or normal saline for 5 days, 2 times a day while keeping current oral anti-parkinsonian medications unchanged
* follow-up after administration of IV amantadine for 4 weeks
* allocation ratio of amantadine:normal saline is 2:1

DETAILED DESCRIPTION:
Intravenous amantadine is known to be effective for parkinsonian motor symptoms abruptly aggravated and for disabling motor symptoms from severe motor fluctuation and dyskinesia in patients with Parkinson's disease. The study investigators experienced several open label cases who were benefit from intravenous amantadine in their parkinsonian motor symptoms and freezing of gait as well. In addition, there is a pilot open label trial in parkinsonian patients with refractory freezing of gait which showed marked benefit in patients with Parkinson's disease, but not in patients with parkinson-plus syndromes.

This study was aimed to evaluate the efficacy of intravenous amantadine in both levodopa-unresponsive freezing of gait and disabling off state freezing of gait in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* the diagnosis of Parkinson's disease according to the United Kingdom Parkinson's Disease Brain Bank criteria
* presence of freezing of gait and the scores of Freezing of Gait Questionnaire 7 or more
* having been treated with oral dopamine replacement therapy for 6 months or more
* score of Korean version of mini-mental status examination is 20 or more

Exclusion Criteria:

* presence of significant cognitive dysfunction, behavioral or psychiatric disorders
* presence of severe cardiac disease
* presence of renal failure, seizure, peptic ulcer disease, liver disease, pheochromocytoma, chronic exhaustive disease, or malignancy
* participation to other clinical trial within 4 weeks
* pregnancy or lactating women
* hypersensitivity to study drugs
* history of intoxication to heavy metals

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
changes in scores on Freezing of Gait Questionnaire | after completion of 5-day schedule of IV amantadine treatment compared with baseline status

SECONDARY OUTCOMES:
changes in scores on Freezing of Gait Questionnaire | after 4-weeks of follow-up compared with baseline status
changes of scores on the Unified Parkinson's disease Rating Scale Part III | after completion of IV amantadine treatment compared with baseline status
changes of scores on the Unified Parkinson Disease Rating Scale Part III | after 4- weeks of follow-up compared with baseline status

CONTACTS AND LOCATIONS:
Overall Officials: Jinwhan Cho, M.D.,Ph.D., Principal Investigator — Department of Neurology, Samsung Medical Center
Locations (4):
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam
  - Hanyang University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul